CLINICAL TRIAL: NCT04115345
Title: A Phase 1 Open-Label Safety, Tolerability, and Early Efficacy Study of a Renal Autologous Cell Therapy (REACT) in Patients With Chronic Kidney Disease From Congenital Anomalies of the Kidney and Urinary Tract (CAKUT) (REGEN-004)
Brief Title: A Study of a Renal Autologous Cell Therapy (REACT) in Patients With Chronic Kidney Disease (CKD) From Congenital Anomalies of the Kidney and Urinary Tract (CAKUT).
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prokidney (Industry)
Collaborators: CTI Clinical Trial and Consulting Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REGEN-004
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-02

CONDITIONS: Chronic Kidney Disease; Congenital Anomalies of Kidney and Urinary Tract
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cakut

STUDY DESIGN:
Intervention Model Description: Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Renal Autologous Cell Therapy (REACT) (Experimental): The volume of REACT to be administered will be determined by pre-procedure MRI volumetric 3D evaluation or ellipsoid formula. The participant will receive a second injection 6 months after the first injection into the same kidney.
  Interventions: Biological: Renal Autologous Cell Therapy (REACT)

INTERVENTIONS:
Biological: Renal Autologous Cell Therapy (REACT) — Autologous selected renal cells (SRC)

SUMMARY:
A phase 1, open-label safety, tolerability and early efficacy study of a Renal Autologous Cell Therapy (REACT) in patients with Chronic Kidney Disease from Congenital Anomalies of the Kidney and Urinary Tract (CAKUT) (REGEN-004)

DETAILED DESCRIPTION:
It is anticipated that all subjects will receive two planned Renal Autologous Cell Therapy (REACT) injections to allow dose-finding and evaluate the duration of effects. The scientific rationale, based on non-clinical studies, is that the biologically active component of REACT (homologous, autologous, SRC) delays progression of experimental models of Chronic Kidney Disease (CKD) by augmenting renal structure and function. As a result, the more cells that can be infused, the greater the potential improvement in renal function.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is male or female, 18 to 65 years of age on the date of informed consent.
2. The patient has a documented history of a corrected abnormality of the kidney and/or urinary tract (CAKUT) leading to renal dysfunction.
3. The patient has an established diagnosis of Stage III/IV CKD not requiring renal dialysis.
4. The subject has blood pressure less than 150/90 at the Screening Visit, prior to renal biopsy, and prior to REACT injection(s).

Exclusion Criteria:

1. The patient has a history of renal transplantation.
2. The patient has a diagnosis of hydronephrosis, SFU Grade 4 or 5.
3. The patient has an uncorrected VUR Grade 5.
4. The patient has a diffuse cortical thickness throughout the kidney measuring < 5 mm on MRI that prevents safe cortical biopsy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Assess change in eGFR and observe incidence of renal-specific procedure and/or product related adverse events (AEs) through 18 months following two Renal Autologous Cell Therapy (REACT) injections [Safety]. | 18 months following last REACT injection
  The primary objective is to assess the safety and optimal delivery of Renal Autologous Cell Therapy (REACT) injected at one site in a recipient kidney as measured by procedure- and/or product related adverse events (AEs) through 18 months post-treatment.

SECONDARY OUTCOMES:
Number of subjects with renal-specific adverse events over a 18-month period following injection of Renal Autologous Cell Therapy (REACT). | 18 months following last REACT injection
  The number of subjects with renal-specific adverse events over a 18-month period following injection of Renal Autologous Cell Therapy (REACT) will be observed utilizing renal-specific laboratory assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Prokidney
Locations (5):
- United States (5):
  - Emory University Hospital, Atlanta, Georgia
  - Boise Kidney & Hypertension Institute, Meridian, Idaho
  - Hackensack Meridian Jersey Shore University Medical Center, Neptune City, New Jersey
  - Mt. Sinai Hospital, New York, New York
  - University of North Carolina- Chapel Hill, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stavas J, Diaz-Gonzalez de Ferris M, Johns A, Jain D, Bertram T. Protocol and Baseline Data on Renal Autologous Cell Therapy Injection in Adults with Chronic Kidney Disease Secondary to Congenital Anomalies of the Kidney and Urinary Tract. Blood Purif. 2021;50(4-5):678-683. doi: 10.1159/000512586. Epub 2021 Mar 1. PMID 33647913